CLINICAL TRIAL: NCT04675736
Title: Evaluation of the Optimum Brushing Force on Dental Plaque Removal and the Abrasive Effect of Brushing Force on Enamel Surface: An in Vitro Study.
Brief Title: Evaluation of the Optimum Brushing Force on Dental Plaque Removal and the Abrasive Effect of Brushing Force on Enamel Surface.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MU-DT/PY-IRB 2017/DT105
Record Dates: First submitted 2020-09-02; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: the Optimum Brushing Force for Dental Plaque Removal and the Effect of Brushing Force on Enamel Characteristic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- brushing force (Experimental)
  Interventions: Procedure: brushing force

INTERVENTIONS:
Procedure: brushing force — Using duplication method, vertical force was applied from 1-5.5 N in linear mesial-distal brushing motion at 4 strokes per second for 5 seconds Force was increase 0.5 N in every testing until plaque was completely removed from enamel surface

SUMMARY:
Objective

1. To determine the optimum brushing force for dental plaque removal.
2. To investigate the effect of brushing force on enamel characteristic.

Hypothesis H0 : Structural tooth loss is not significantly different between before and after brushing with excessive force on enamel surface.

H1 : Structural tooth loss is significantly different between before and after brushing with excessive force on enamel surface.

Study design: Experimental study

ELIGIBILITY:
Inclusion Criteria:

* extracted bovine incisors

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
optimum force | 5 seconds
  The toothbrush holder was adjusted allowing toothbrush bristle to press onto the tooth surface until the loading monitor indicated the designated vertical loading force. Loading force was applied from a minimum of 1 N, with an increment of 1 N to a maximum of 6 N. The optimum force which remove all dental plaque from tooth surface will recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Kanyawat rattanasuwan, Study Director — Department of Oral Medicine and Periodontology, Faculty of Dentistry, Mahidol University, Bangkok Thailand
Locations (1):
- Faculty of Dentistry, Ratchathewi, Bangkok, Thailand